CLINICAL TRIAL: NCT05071924
Title: Parenting for Lifelong Health for Teens - Hybrid Delivery
Brief Title: PLH for Teens - Hybrid Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mothers2Mothers (Unknown); University of Cape Town (Other)
Responsible Party: Principal Investigator, DrJamieLachman, Principal Investigator, University of Oxford
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PLH/M2M/HY21
Record Dates: First submitted 2021-09-27; First posted 2021-10-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Child Maltreatment; Positive Parenting
Keywords: Parenting programme; Child physical and emotional abuse

STUDY DESIGN:
Intervention Model Description: This is a pre-post study with assessments at baseline and immediate post- intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLH Teens Original (Experimental): The original in-person PLH programme is delivered by community-based workers in low-resource settings. Implementation occurs in a group-based format with both joint parent and teen sessions (10 sessions) and separate parent and teen sessions (4 sessions).
  Interventions: Behavioral: PLH Teens Original: In-person PLH programme for parents and teens by community-based workers
- PLH Teens Hybrid (Experimental): The hybrid delivery of PLH Teens consists of 8 sessions delivered to parents via WhatsApp (ParentChat-Teens) and 4 sessions delivered to parents and adolescents in person.
  Interventions: Behavioral: PLH Teens Hybrid: Hybrid delivery for parents and teens by facilitators

INTERVENTIONS:
Behavioral: PLH Teens Original: In-person PLH programme for parents and teens by community-based workers — This in-person intervention is delivered over 14 sessions (10 joint parent and teen sessions and 4 separate parent and teen sessions).
  Arms: PLH Teens Original
Behavioral: PLH Teens Hybrid: Hybrid delivery for parents and teens by facilitators — The hybrid intervention delivered over 12 sessions (8 sessions delivered via WhatsApp groups to parents only and 4 sessions delivered in-person to parents and teens together).
  Arms: PLH Teens Hybrid

SUMMARY:
This study aims to examine the implementation and effectiveness of the original version of PLH Teens delivered in-person (PLH Teens-Original) and a hybrid in-person and remote delivery of the programme (PLH Teens-Hybrid) as part of the Mothers2Mothers' (M2M) Children and Adolescents are My Priority (CHAMP) project in Mpumalanga, South Africa. It will also examine differential effects between PLH Teens-Original and PLH Teens-Hybrid on reducing risks of violence against children using propensity score matching. Lastly, it will examine the implementation feasibility of PLH Teens-Hybrid in terms of implementation fidelity; recruitment, retention, and engagement of parents and adolescents; and the relevance, acceptability, and satisfaction of the programme.

DETAILED DESCRIPTION:
Study Design This study will use a mixed-methods approach to qualitatively and quantitatively address the research aims. It will be implemented from May to July 2021 in the Mpumalanga province of South Africa. The study design will involve a) pre-post quantitative analyses of primary and secondary outcomes for both PLH Teens-Original and PLH Teens-Hybrid, b) difference in analyses to compare effects between the two delivery modalities, and c) qualitative interviews and quantitative analyses of programme feasibility and implementation.

Recruitment Recruitment of parents/caregivers and adolescents will be integrated into CHAMP's current recruitment strategy which includes engaging with schools, faith-based organisations, local NGOs, health facilities, United States Agency for International Development (USAID) DREAMS (Determined, Resilient, Empowered, AIDS-free, Mentored, and Safe) partners, door-to-door engagement and other contextually relevant approaches. CHAMP leverages its partnerships for recruitment and the CHAMP partner, Grassroots Soccer, actively engages in recruitment for the DREAMS programme. Participants enrolled into the hybrid PLH programme will be screened using the USAID approved Vulnerability Assessment Tool to ensure that the most vulnerable households are reached. The pilot will target caregivers in the Nelspruit area to ensure adequate access to internet connectivity.

ELIGIBILITY:
Inclusion criteria for participating parents or caregivers:

* Any person over the age of 18 currently caring for a child between the ages of 10 and 17
* Has the ability to attend the in-person parenting support group (PLH Teens-Original)
* Has access to a WhatsApp compatible smartphone and is willing to join an online parenting support group (PLH Teens-Hybrid)
* Has provided consent to participate in the study

Inclusion criteria for teens:

* Must be between the age of 10 and 17
* Has a parent or caregiver who is participating in the programme
* Parent has provided consent to participate in the study
* Has provided assent to participate in the study

Inclusion criteria for facilitators:

* The facilitator must be over the age of 18
* Has completed a facilitator training workshop specifically for the PLH-Teens hybrid delivery prior to intervention delivery
* Is able to access the in-person session location
* Has a smart-phone or device capable of delivering the programme via an online platform such as WhatsApp or Viber
* Has provided informed consent to participate in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1128 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Child Maltreatment: ISPCAN Child Abuse Screening Tools-Trial Version - Parent Report | Change between Baseline and Post (approx. 4 months post-baseline)
  Child maltreatment will be assessed using a shortened version of the ISPCAN Child Abuse Screening Tools-Trial Version (9-item subscale ICAST-T). Parent respondents will be asked to indicate the frequency of emotional and physical discipline practices over the past month using a 9-point frequency count scale (0 = never; 8 = 8 or more times). Items include, "In the past 4 weeks, how often did you/your caregiver discipline your child/you by spanking, slapping or hitting with a hand?" and "In the past 4 weeks, how often did you/your caregiver shout, yell or scream at you?" In the past 4 weeks, how often did you/your caregiver discipline your child/you with an object like a stick or a belt?". Items are summed, with higher scores indicating greater use of harsh parenting.
Child Maltreatment: ISPCAN Child Abuse Screening Tools-Trial Version - Teen Report | Change between Baseline and Post (approx. 4 months post-baseline)
  Child maltreatment will be assessed using a shortened version of the ISPCAN Child Abuse Screening Tools-Trial Version (9-item subscale ICAST-T). Teen respondents will be asked to indicate the frequency of emotional and physical discipline practices over the past month using a 9-point frequency count scale (0 = never; 8 = 8 or more times). Items include, "In the past 4 weeks, how often did you/your caregiver discipline your child/you by spanking, slapping or hitting with a hand?" and "In the past 4 weeks, how often did you/your caregiver shout, yell or scream at you?" In the past 4 weeks, how often did you/your caregiver discipline your child/you with an object like a stick or a belt?". Items are summed, with higher scores indicating greater use of harsh parenting.

SECONDARY OUTCOMES:
Parenting Stress: Parenting Stress Scale | Change between Baseline and Post (approx. 4 months post-baseline)
  Parenting Stress will be assessed using the Parenting Stress Scale (7-item PSS subscale; Berry & Jones, 1995). The PSS asks parents to respond to items related to positive (e.g., "I feel close to my child") and negative (e.g., "I feel overwhelmed by the responsibility of being a parent") feelings related to parenting stress using a 5-point Likert-like scale (1 = Strongly disagree; 5 = Strongly agree). After reverse-coding certain items, items will be summed with higher scores indicating higher levels of parenting stress.
Child Maltreatment - Physical Abuse and Emotional Abuse: ISPCAN Child Abuse Screening Tool-Intervention (ICASTTP) - Physical and Emotional Abuse Subscales | Change between Baseline and Post (approx. 4 months post-baseline)
  Physical abuse and emotional abuse will be measured using 4 items from a reduced version of the ISPCAN Child Abuse Screening Tool-Trial Parent version (ICAST-TP). The ICAST-TP measures parental reports of the incidence of abuse perpetrated against their child over the past month using a frequency score on a scale of 0 to 7, or 8 or more times (e.g., "In the past 4 weeks, how often did you discipline your child by spanking, slapping, or hitting with your hand?").
Positive Parenting: Alabama Parenting Questionnaire - Parent Report | Change between Baseline and Post (approx. 4 months post-baseline)
  Positive parenting will be assessed based on parent-report of an adapted version of the Alabama Parenting Questionnaire (6-item APQ subscale; Frick, 1991). The APQ measures the frequency of specific behaviours towards children in the past month on a 7-point Likert-like scale (e.g., "You talk to your child about their friends"; 0 = never; 6 = always). Items are summed to create a frequency score, with higher scores indicating more regular use of positive parenting.
Positive Parenting: Alabama Parenting Questionnaire - Teen Report | Change between Baseline and Post (approx. 4 months post-baseline)
  Positive parenting will be assessed based on teen-report of an adapted version of the Alabama Parenting Questionnaire (6-item APQ subscale; Frick, 1991). The APQ measures the frequency of specific behaviours towards children in the past month on a 7-point Likert-like scale (e.g., "Your caregiver talks to you about your friends"; 0 = never; 6 = always). Items are summed to create a frequency score, with higher scores indicating more regular use of positive parenting.
Child Behaviour Problems: Strengths and Difficulties Questionnaire - Parent Report | Change between Baseline and Post (approx. 4 months post-baseline)
  Child behaviour problems will be assessed using parent-report of the Strengths and Difficulties Questionnaire (10-item SDQ; Goodman, 1997). Respondents will be asked to report on the frequency of specific child behaviours (e.g., "Your child is restless, overactive, cannot stay still for long" using a 3-point Likert-like scale (1 = Not true; 3 = Very true). Items are summed, with higher scores indicating more behavioural problems.
Child Behaviour Problems: Strengths and Difficulties Questionnaire - Teen Report | Change between Baseline and Post (approx. 4 months post-baseline)
  Child behaviour problems will be assessed using teen-report of the Strengths and Difficulties Questionnaire (10-item SDQ; Goodman, 1997). Respondents will be asked to report on the frequency of specific child behaviours (e.g., "You are restless, overactive, cannot stay still for long" using a 3-point Likert-like scale (1 = Not true; 3 = Very true). Items are summed, with higher scores indicating more behavioural problems.
Parental Depression: Centre for Epidemiologic Studies Depression Scale - Parent Report | Change between Baseline and Post (approx. 4 months post-baseline)
  Parental depression will be assessed using the Centre for Epidemiologic Studies Depression Scale (10-item CES-D subscale; Radloff, 1977). Caregivers will be asked to respond to items related to how they have felt over the past seven days (e.g., "How often in the past week have you been bothered by things that don't usually bother you?"). Responses are coded on a 4-point Likert-like scale (i.e., 1 = Rarely or none of the time (less than 1 day) to 4 = Most or all of the time (5 to 7 days)) and summed to create a total of parental depression.
Teens Internalising Behaviours: Strength and Difficulties Questionnaire (SDQ) - Parent Report | Change between Baseline and Post (approx. 4 months post-baseline)
  Teen internalising behaviours will be assessed using parent-report of the Strengths and Difficulties Questionnaire (SDQ) based subscales for emotional problems (e.g. "I worry a lot") and peer problems (e.g. "I am usually on my own. I generally play alone or keep to myself") (15-item SDQ subscale; Goodman, 1997). Items are summed to create a total measurement of internalising behaviour.
Risk Avoidance: Risk Avoidance Planning Scale - Parent Report | Change between Baseline and Post (approx. 4 months post-baseline)
  Risk Avoidance will be assessed using parent-report of the Risk Avoidance Planning Scale (5-item RAPS; Cluver et al., 2018). Caregivers will be asked whether they have spoken to their child about risks in the community including topics such as safe sex and community safety. This scale was developed specifically for the PLH for Teens programme in South Africa (Cluver et al., 2018). Caregivers will be asked to respond on a 3-point Likert-like scale as to whether they have spoken to their child about risks in the community (1 = No, I find it too hard to talk about this; 2 = We haven't made plans yet but I would like to talk about it; 3 = We have made a plan together). Topics will include safe sex and community safety.
Risk Avoidance: Risk Avoidance Planning Scale - Teen Report | Change between Baseline and Post (approx. 4 months post-baseline)
  Risk Avoidance will be assessed using teen-report of the Risk Avoidance Planning Scale (5-item RAPS; Cluver et al., 2018). Teens will be asked to respond on a 3-point Likert-like scale as to whether they have spoken about risks in the community (1 = No, I find it too hard to talk about this; 2= We haven't made plans yet but I would like to talk about it; 3 = We have made a plan together). Topics will include safe sex and community safety.
Economic Strengthening: Family Financial Coping Scale - Parent Report | Change between Baseline and Post (approx. 4 months post-baseline)
  Economic Strengthening will be measured using a Family Financial Coping Scale (5-item FFCS; Lown, 2011). Caregivers will be asked to respond to household demographic items over the past month. These items cover a variety of financial matters including whether caregivers were worried about money, whether they managed to save money, and whether they ran out of money to buy certain items, including food, transport, and mobile data or airtime. Responses are coded on a 4-point Likert scale (0 = Never, 1 = Rarely, 2 = Sometimes, 3= Often). Items are summed, with a higher score reflected a greater number of financial challenges.
Economic Strengthening: Family Financial Coping Scale - Teen Report | Change between Baseline and Post (approx. 4 months post-baseline)
  Economic Strengthening will be measured using a Family Financial Coping Scale (5-item FFCS; Lown, 2011). Teens will be asked to respond to household demographic items over the past month. These items cover a variety of financial matters including whether caregivers were worried about money, whether they managed to save money, and whether they ran out of money to buy certain items, including food, transport, and mobile data or airtime. Responses are coded on a 4-point Likert scale (0 = Never, 1 = Rarely, 2 = Sometimes, 3= Often). Items are summed, with a higher score reflected a greater number of financial challenges.
Parent Support of Education: Parental Support for School Scale - Parent Report | Change between Baseline and Post (approx. 4 months post-baseline)
  Parent Support of Education will be measured using an adapted version of the Parental Support for School Scale (6-item PSE; Ceballo, Maurizi, Suarez, & Aretakis, 2014). Caregivers will report on the frequency of supportive behaviour towards children's learning (e.g. "I support my child's schoolwork in any way that I can" and "I praise my child for working hard at school") using a 5-point Likert-like scale (1 = never; 5 = always). Items are summed to create a frequency score, with higher scores suggesting more parental support and value for school. Items from this survey are present in both the parent survey.
Parent Support of Education: Parental Support for School Scale - Teen Report | Change between Baseline and Post (approx. 4 months post-baseline)
  Parent Support of Education will be measured using an adapted version of the Parental Support for School Scale (6-item PSE; Ceballo, Maurizi, Suarez, & Aretakis, 2014). Teens will report on the frequency of supportive behaviour towards children's learning (e.g. "support your schoolwork in any way that he/she can" and "praise you for working hard at school") using a 5-point Likert-like scale (1 = never; 5 = always). Items are summed to create a frequency score, with higher scores suggesting more parental support and value for school. Items from this survey are present in the teen survey.
Attitude Toward Punishment: UNICEF Multiple Indicator Cluster Survey (MICS) 5 Child Discipline Module - Teen Report | Change between Baseline and Post (approx. 4 months post-baseline)
  Attitude toward punishment will be measured using a single-item from the UNICEF Multiple Indicator Cluster Survey (MICS) 5 Child Discipline module - Teen Report (1-item; ). Teens will be asked to report on whether they agree or disagree with the statement: "In order to bring up, raise up, or educate a child properly, the child needs to be physically punished".
Attitude Toward Punishment: UNICEF Multiple Indicator Cluster Survey (MICS) 5 Child Discipline Module - Parent Report | Change between Baseline and Post (approx. 4 months post-baseline)
  Attitude toward punishment will be measured using a single-item from the UNICEF Multiple Indicator Cluster Survey (MICS) 5 Child Discipline module - Teen Report (1-item; ). Caregivers will be asked to report on whether they agree or disagree with the statement: "In order to bring up, raise up, or educate a child properly, the child needs to be physically punished".

OTHER OUTCOMES:
Demographics: Demographic Survey - Parent Report | Baseline
  Basic demographic information will be collected at baseline and post-test for caregivers. Demographic information will include; age, gender, literacy, family structure and dynamics, and risk behaviours. During screening family risk will also be assessed using a Vulnerability assessment tool as a proxy assessment of vulnerability to understand the socio-economic needs of respondents (USAID, 2012). There are six questions that will be asked to respondents which are drawn from the topic of child protection, access to education, nutrition status, child's care and support, child social behaviour, and access to health. Each question will either be in a form of Likert or multiple choice question and have a maximum score of 4. Higher total score indicates lower vulnerability.
Demographics: Demographic Survey - Teen Report | Baseline
  Basic demographic information will be collected at baseline and post-test for teens. Demographic information will include; age, gender, literacy, family structure and dynamics, and risk behaviours. During screening family risk will also be assessed using a Vulnerability assessment tool as a proxy assessment of vulnerability to understand the socio-economic needs of respondents (USAID, 2012). There are six questions that will be asked to respondents which are drawn from the topic of child protection, access to education, nutrition status, child's care and support, child social behaviour, and access to health. Each question will either be in a form of Likert or multiple choice question and have a maximum score of 4. Higher total score indicates lower vulnerability.
Enrolment Rates of Participant Engagement: Weekly Facilitator Survey - Facilitator Report | Weekly from week 1- 12 for hybrid delivery and week 1-14 for in-person delivery
  Facilitator programme adherence will be assessed by examining rates of enrolment.
Attendance Rates of Participant Engagement: Weekly Facilitator Survey - Facilitator Report | Weekly from week 1- 12 for hybrid delivery and week 1-14 for in-person delivery
  Facilitator programme adherence will be assessed by examining rates of attendance.
Dropout Rates of Participant Engagement: Weekly Facilitator Survey - Facilitator Report | Weekly from week 1- 12 for hybrid delivery and week 1-14 for in-person delivery
  Facilitator programme adherence will be assessed by examining rates of dropout. Dropout rates for enrolled participants will be defined as the percentage of participants who do not attend at least two consecutive sessions across either the in-person or online components of the programme, and do not attend any sessions at a later stage.
Implementation Fidelity: Facilitator Report | Weekly from week 1- 12 for hybrid delivery and week 1-14 for in-person delivery
  Implementation fidelity of the hybrid PLH programme will be measured using self-report checklists by facilitators to understand the extent to which core intervention components are delivered. These checklists will include specific activities for each session in both the in-person and at home components of the programme. Then, in order to produce a basic level of fidelity, a ratio of programme implementation to programme design will be created for the self-report scores. A score of 80% programme fidelity will be considered as "high treatment fidelity".
Intervention Cost of Programme for Scale-up: Facilitator Report | Weekly from week 1- 12 for hybrid delivery and week 1-14 for in-person delivery
  Intervention cost of programme for scale-up will be assessed using facilitator reports of the time and resource costs spent delivering the programme. This will include training and preparation for delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie M. Lachman, DPhil, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be shared on Open Science Framework after the completion of the study and results are published.
Supporting Information: Study Protocol
Time Frame: Indefinitely
Access Criteria: Accessibility of the data will require approval from the study team. The study investigators, led by the PI, will jointly make decisions on whether to supply research data to potential new users. Research data will be deposited in and available in the UK Data Archive solely for non-profit use.